CLINICAL TRIAL: NCT02507037
Title: Effect of Gum Chewing on Bowel Cleansing Before Colonoscopy: A Prospective Randomized Study
Brief Title: Effect of Gum Chewing on Bowel Cleansing Before Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept., Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Gum-1
Record Dates: First submitted 2015-07-19; First posted 2015-07-23 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Bowel Preparation Scale; Adenoma Detection Rate
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gum+PEG (Experimental): used 2L PEG+sugarless gum
  Interventions: Dietary Supplement: gum+PEG
- PEG (Placebo Comparator): only used 2L PEG
  Interventions: Drug: polyethylene glycol

INTERVENTIONS:
Dietary Supplement: gum+PEG — chew sugarless gum
  Arms: gum+PEG
Drug: polyethylene glycol — 2L PEG
  Arms: PEG

SUMMARY:
In this randomized controlled study, consecutive outpatients scheduled for elective colonoscopy were randomized into two groups. Group A patients (n = 150) used 2 L PEG before colonoscopy. Patients in group B (n = 150) were additionally advised to chew sugarless gum plus 2 L PEG, The overall quality of colonoscopy cleaning was evaluated using the Boston Bowel Preparation Scale by endoscopists who was blinded to the intervention. Difficulty of procedure, patients' tolerance, and adverse events were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All adults (18-65) who were referred for outpatient colonoscopy.

Exclusion Criteria:

* under 18 years or More than 65 years
* previous abdominal surgery
* major psychiatric disorders
* pregnancy
* presence of any contraindications for colonoscopy(eg, severe heart failure)
* recent inadequate colonoscopy history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | 2 days

SECONDARY OUTCOMES:
number of patient tolerability | 2 days
number of patient willingness to repeat preparation | 2 days
Adenoma Detection Rate | 2 days

REFERENCES:
- [Result] Sakin YS, Uygun A, Bagci S. Comment on: Efficacy and safety of gum chewing in adjunct to high-dose senna for bowel cleansing before colonoscopy: a single-blind randomized controlled trial. Saudi J Gastroenterol. 2015 Jan-Feb;21(1):56. doi: 10.4103/1319-3767.151233. No abstract available. PMID 25672242
- [Result] Ergul B, Filik L, Kocak E, Dogan Z, Sarikaya M. Efficacy and safety of gum chewing in adjunct to high-dose senna for bowel cleansing before colonoscopy: a single-blind randomized controlled trial. Saudi J Gastroenterol. 2014 Nov-Dec;20(6):356-9. doi: 10.4103/1319-3767.145325. PMID 25434316
- [Result] Ou G, Svarta S, Chan C, Galorport C, Qian H, Enns R. The effect of chewing gum on small-bowel transit time in capsule endoscopy: a prospective, randomized trial. Gastrointest Endosc. 2014 Apr;79(4):630-6. doi: 10.1016/j.gie.2013.08.038. Epub 2013 Oct 7. PMID 24112594
- [Derived] Fang J, Wang SL, Fu HY, Li ZS, Bai Y. Impact of gum chewing on the quality of bowel preparation for colonoscopy: an endoscopist-blinded, randomized controlled trial. Gastrointest Endosc. 2017 Jul;86(1):187-191. doi: 10.1016/j.gie.2016.05.051. Epub 2016 Jun 17. PMID 27327849